CLINICAL TRIAL: NCT01087450
Title: The Effect of rHuEPO on Microcircualtory Alteration in ICU Patients With Severre Sepsis and Septic Shock
Brief Title: The Effect of Erythropietin on Microcircualtory Alteration in Intensive Care Unit Patients With Severe Sepsis
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Raymond Kao, Physician, London Health Sciences Centre
Other Study IDs: 15474
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Sepsis; Shock
Keywords: Erythropoietin; Sepsis; Septic shock; Orthogonal Polarization Spectroscopy; Severe sepsis or Septic shock
MeSH Terms: conditions — Sepsis; Shock; Shock, Septic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stage1: 1. Prospective dose response group. 3 subjects per dose at 200U/kg, 400U/kg and 600U/kg rHuEPO
- Stage 2 Randomized, blinded trial: Control group: Randomized to placebo treatment Treatment Group: Randomized to rHuEPO treatment

SUMMARY:
The objective of this study is to determine if observations the investigators made in an animal model of sepsis can be translated to clinical practice. Specifically, the investigators will use the noninvasive Orthogonal Polarization Spectral (OPS) microscope and venous oxygen saturation to test the hypothesis that recombinant human erythropoietin(rHuEPO) will acutely improve the microcircualtion in septic patients in the ICU.

DETAILED DESCRIPTION:
Sepsis is a systemic inflammatory response to a bacterial infection and is a common complication during the course of treatment of patients with multiple trauma and major surgery. In severe sepsis, the inflammatory response leads to multiple organ failure that can result in death. Multiple organ dysfunction in sepsis is now considered the most common cause of death in non-coronary critical care units. In fact, sepsis is one of the top 10 or 12 causes of death in the general population. Approximately 150,000 people die annually.1 On a microscopic level there is impairment in the relationship between oxygen delivery (DO2) and consumption (VO2) suggestive of defects in microcirculatory perfusion during septic shock.2,3,4 These alterations include a decrease in the proportion of perfused vessels smaller than 20 μm, which mostly are capillaries whereas flow in the larger perfusion vessels is preserved. As the micro-circulation alteration persists then multiple organ failure and death ensues,4 thus interventions able to improve the microcirculation may reduce tissue dysoxia. De Backer et. al.3 reported that topical application of acetylcholine can restore a normal microcirculatory flow pattern in patients with septic shock, indicating an important role for the micro-vascular endothelium, and that these alterations can be manipulated. Other experimental studies of several vasodilatory compounds have been shown to improve micro-vascular perfusion5,6,7,8,9 and even be associated with improved outcomes.7,10 In a human study, Spronk et. al.11 observed that intravenous administration of nitroglycerin resulted in a marked improvement in capillary perfusion, but this intervention may produce severe arterial hypotension and also increase some nitric oxide mediated cytoxic effects.12,13 In another human study, De Baker et. al.14 demonstrated that the administration of 5 μg/kg-min dobutamine can improve but not restore capillary perfusion in patients with septic shock and that these changes are independent of changes in systemic hemodynamic variables. The concomitant decrease in blood lactate level suggested the changes in the micro-vascular perfusion were associated with improved cellular metabolism. However, dobutamine may also produce hypotension in patients with hypovolemia.

Erythropoietin (EPO), a sialoglycoprotein hormone produced by the adult kidney, is a major regulator of red blood cell production but more recently has been suggested to have favourable effects on tissue injury and vascular function. It stimulates the proliferation of committed erythroid progenitor cells and their development into mature erythrocytes.15 Thus, the potential benefit of erythropoietin therapy in patients with anemia secondary to chronic renal failure has long been recognized.16 Recombinant Human EPO (rh-EPO) is indicated for the treatment of anemia associated with chronic renal failure, non-myeloid malignancies due to the effect of concomitantly administered chemotherapy, zidovudine treated HIV infected patients and patients under going major elective surgery to facilitate autologous blood collection thus to reduce allogenic blood exposure.

In critically ill adults and specifically those with sepsis, EPO levels have been shown to be relatively low with respect to the level of anemia present.17,18 As well, correlations were found between erythropoietin concentration and biological markers of tissue hypoperfusion i.e. lactate level or PCO2 gap.19 A common adverse effect of rh-EPO therapy in renal patients is the development of hypertension. The acute effects of rh-EPO on arterial vasoactivity suggest direct and indirect actions that occur prior to any effect on erythropoeisis. In addition to its hematopoietic effect, rh-EPO also has significant cardiovascular effects,20,21 including a direct vasopressor effect.22 In a rat splanchnic artery occlusion shock model, treatment with rh-EPO inhibited inducible nitric oxide synthase (iNOS) activity and prevented the overproduction of NO in vivo restoring responsiveness to Phenylephrine.23,24 Rh-EPO has direct vasopressor effects on smooth muscle cells, which express EPO receptors, modulating intracellular Ca++.25 An increase in the plasma levels of the endothelium derived vasoconstrictor endothelin-1 can occur after rh-EPO treatment.26,27,28 Indirect effects of EPO treatment may also increase the activity of the autonomic nervous system and increase sensitivity to angiotensin II, which is a potent vasoconstrictor.29 We recently reported that rh-EPO in a septic mouse model produces an immediate increase in the perfused capillary density with a concomitant decrease in NADH fluorescence, an indirect measure indicating improvement in mitochondical oxidative phosphorylation, in skeletal muscle. Thus, rh-EPO appears to improve tissue bioenergetics in this septic mouse model in part by maintaining DO2 via increased perfused capillary density.30 The recently developed, noninvasive orthogonal polarization spectral (OPS) imaging technique can be applied to investigate the human vasculature.34 Polarized light of defined wavelength (548 nm) is emitted to illuminate the area of interest, is reflected by the background but absorbed by hemoglobin, producing high-contrast images of the micro-circulation. This technique is particularly convenient for studying tissues protected by a thin epithelial layer, such as the mucosal surface35 and has been validated as an effective method of micro-vascular imaging in animals34, 36,37 and in humans.38 The OPS technique has been used to observe major micro-vascular blood flow alterations in patients with severe sepsis3 including a decreased vascular density, especially of the small vessels; a large number of non-perfused and intermittently perfused small vessels; and a marked perfusion heterogeneity between areas.39 These alterations were more severe in non-survivors than in survivors but were not affected by the global hemodynamic state or vasopressor agents.39 The persistence of micro-vascular alterations in patients with poor outcomes further emphasize the potential role of micro-circulatory disturbances in the pathophysiology of sepsis-induced multiple organ failure. In this study, we will use the OPS imaging technique to investigate the sublingual microcirculation in patients with septic shock after treatment with a single dose of rh-EPO. We hypothesize that rh-EPO will improve the sepsis-related alterations in micro-circulatory perfusion, independent of any systemic hemodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* The patients must be 18 years old and over to be included in the study. They must meet criteria for sepsis defined as:40

  1. Two or more criteria for the systemic inflammatory response syndrome (SIRS):

     * heart rate greater than 90 beats per minute, or paced, or taking beta-blockers or the calcium channel blockers verapamil or diltiazem
     * respiratory rate greater than 20 breathes per minute, or a PaC02 less than 32 mmHg, or mechanically ventilated
     * temperature greater than 38 or less than 36 degrees Celsius
     * white blood cell count greater than 12 x 109/L or less than 4 x 109/L, or more than 10% bands on the differential.
  2. Suspected or confirmed source of infection

     And either one of the following definitions:
  3. Severe Sepsis: Sepsis with at least one organ dysfunction defined as urine output < 0.5 ml/kg/hr for 1 hour, PaO2/FiO2 < 250 (less than 200 if lung is the only dysfunctional organ), platelets < 80 x109/L or a 50% decrease from baseline in the past 3 days, or pH < 7.30 or lactate > 1.5 mmole/L upper normal with base deficit > 5
  4. Septic shock <48hrs: Persistent arterial hypotension with a systolic pressure < 90 mmHg or a MAP < 60 mmHg or a reduction of in systolic blood pressure > 40 mmHg from baseline, despite adequate fluid resuscitation in the absence of other cause for hypotension or requiring the administration of a pressor agent to maintain the above blood pressure.

Exclusion Criteria:

* Clinically apparent other forms of shock including cardiogenic, obstructive (massive pulmonary embolism, cardiac tamponade, tension pneumothorax) or hemorrhagic shock
* A known previous severe reaction to erythropoietin
* Uncontrolled hypertension (hypertensive urgency, hypertensive emergency and hypertensive encephalopathy)
* Myocardial infarction and/or stroke within one month
* Hypersensitivity reaction after previous rh-EPO use. Known sensitivity to products from mammalian cell cultures
* Previous history of deep venous thromboses or pulmonary embolism
* Burns
* Cirrhosis
* Traumatic brain injury
* Less than 18 years of age
* Family or patient not committed to aggressive care
* Currently enrolled in another related interventional study
* Any active cancer patients of any type and stage except for patients with basal and squamous cell skin cancers
* Patient weighing > 100 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment Critical Care research coordinators and a Research Fellow will screen patients for severe sepsis and septic shock in the London Health Sciences Center-Critical Care Trauma Center (LHSC-CCTC). The patients who meet the inclusion criteria will be introduced to this study. Informed consent will be obtained from the patient or a family member or a substitute decision maker.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-08-12 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Changes in sub-lingual micro-circulatory blood flow for each enrolled subject using the Orthogonal Polarization Spectral imaging at three time points | 1. Baseline; 2. At 1-hour post treatment with EPO or placebo; 3. At 24-hours post treatment with EPO or placebo
  1. Semi-quantitative analysis on all images off-line for microcirculatory flow characteristics the units utilized is Percent Perfused Vessel analysis (PPV%)
  2. It is proposed that with improved PPV% there will be improved venous blood and tissue oxygen saturation.

SECONDARY OUTCOMES:
1. Changes in splanchnic venous oxygen saturation at three time points for each subject. 2. Changes in tissue oxygen saturation of the thenar eminence muscle at three time points for each subject. | 1. At baseline 2. 1- hour post treatment or placebo 3. At 24 hors post treatment or placebo
  1. Utilizing the blood gas machine in the Intensive Care Unit to measure the splanchnic venous oxygen saturation (SpVo2 or percent saturation) from the venous blood drawn from the femoral central venous catheter.
  2. Utilizing the In-Spectra monitor model 650 to measure the thenar eminence muscle tissue oxygen saturation or percent saturation.
  3. With an improvement of microcirculation in the sub-lingual region there should also be oxygenation saturation improvement in the splanchnic blood pool region and tissue oxygen saturation improvement in the thenar eminence muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Center-Critical Care Trauma Center, London, Ontario, Canada